CLINICAL TRIAL: NCT03219320
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multiple-Dose Study to Assess the Efficacy and Safety of NYX-2925 in Subjects With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Efficacy and Safety of NYX-2925 in Subjects With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Acronym: DPN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NYX-2925-2001
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Type 2 Diabetes; Neuropathic Pain; Peripheral Nervous System
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuralgia | interventions — NYX-2925

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive placebo or NYX-2925.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment arms, dose levels, and randomization algorithm are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Oral Capsule (Placebo Comparator): Up to 300 subjects: Placebo
  Interventions: Drug: Placebo
- NYX-2925 (Experimental): Up to 300 subjects: Multiple dose levels of NYX-2925 daily for 28 days
  Interventions: Drug: NYX-2925

INTERVENTIONS:
Drug: NYX-2925 — NYX-2925 is a novel small molecule that modulates the N-methyl-D-aspartate receptor (NMDAR).
  Arms: NYX-2925
Drug: Placebo — Matching Placebo capsules.
  Arms: Placebo Oral Capsule

SUMMARY:
To evaluate the efficacy of multiple dose levels of NYX-2925 versus placebo in treating the neuropathic pain associated with Diabetic Peripheral Neuropathy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, placebo-controlled, multiple-dose study to assess the efficacy and safety of NYX-2925 in subjects with neuropathic pain associated with diabetic peripheral neuropathy.

The study will be a 6 to 9-week study, including a 1 to 4-week (dependent on duration of washout period) Screening Period, followed by a 4-week double-blind, randomized, placebo-controlled Treatment Period, and a 1-week Follow Up Period. Subjects eligible for the study will randomize to receive either NYX-2925 or placebo for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board-approved written informed consent and privacy language (Health Insurance Portability and Accountability Act) authorization must be obtained from the subject prior to performing any study-related procedures.
2. Subjects who consent to being included in a subject registry database.
3. Male and female subjects ≥18 and ≤75 years of age.
4. Subjects with a diagnosis of Type 2 diabetes.
5. Subjects with a score of ≥4 and ≤9 on the 11-point numeric rating scale (NRS) for average pain intensity over the past 24 hours at Visit 1.
6. Hemoglobin A1c (HbA1c) ≤11% (measured at Visit 1).
7. Stable use of diabetic medications beginning 1 month prior to Visit 1 (Adequate glycemic control with only diet and exercise is also permitted.).
8. Subjects with diabetic peripheral neuropathy, of symmetrical nature and in lower extremities for ≥6 months to ≤10 years, and diagnosed by a score of ≥3 on Michigan Neuropathy Screening Instrument.
9. Body mass index of <40 kg/m^2
10. Calculated creatinine clearance of ≥60 mL/minute (Cockcroft-Gault formula).
11. Clinical laboratory values must be within normal limits or deemed not clinically significant by the investigator and sponsor-designated medical monitor.

Inclusion Criteria: Randomization Daily pain scores and diary compliance will be transferred into the interactive response technology system, which will assess the criteria for randomization. Subjects whose mean of the daily average pain intensity score during the preceding 7 (±1) days is within the protocol-defined algorithm and with adequate compliance with daily diary completion will be eligible for randomization.

Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

1. Subjects who have a current diagnosis of major psychiatric disorder (including schizophrenia, bipolar disorder, or panic disorder), including those who have required an antipsychotic or mood stabilizer (e.g., lithium, carbamazepine, valproate) for a psychiatric condition in the past year, or subjects who have had a major depressive episode (MDE) in the past 6 months. Subjects with major depressive disorder (MDD) or generalized anxiety disorder (GAD) who have been on stable medications for the past 3 months (and are expected to remain stable for the duration of the trial) and whose condition is currently well-controlled may be included.
2. Subjects who have pain that cannot be clearly differentiated from, or could interfere with the assessment of peripheral diabetic neuropathy, as measured by the Masquerading Disorders Tool at Visit 1.
3. Neurologic disorders unrelated to diabetic neuropathy (e.g., phantom limb from amputation), skin condition in the area of neuropathy that could alter sensation (e.g., plantar ulcer), or other painful conditions (e.g., arthritis) that, in the judgment of the investigators, could interfere with reporting of pain due to diabetic neuropathy.
4. History of hypoglycemia that disturbed consciousness, or ketoacidosis requiring hospitalization within past 3 months.
5. Subjects with history of severe renal impairment.
6. Impaired hepatic function.
7. Known history of significant cardiovascular condition.
8. History of Huntington's disease, Parkinson's disease, Alzheimer's disease, Multiple Sclerosis, or a history of seizures, epilepsy, or strokes.
9. HIV infection, hepatitis, or other ongoing infectious disease that the investigator considers clinically significant.
10. Concomitant use of antiepileptic drugs, non-steroidal anti-inflammatory drugs (except cardiac preventive acetylsalicylic acid), opioids, muscle relaxants, dextromethorphan (except low dose intermittent use for cough), tramadol, topical lidocaine, topical capsaicin, and selective norepinephrine reuptake inhibitors. Subjects are allowed to enter with a maximum of 1 allowed analgesic medication for neuropathic pain that has been taken at stable dose for at least 1 month (30 days) prior to Visit 1. Allowed analgesics may not be N-methyl-D-aspartate receptor ligands, must be non-opioid and non-sedative and must not interfere with subjects' pain reporting. Tricyclic antidepressants may be continued if designated as the single analgesic medication for the treatment of pain.
11. Sensitivity to, allergy to, or concomitant use of N-methyl-D-aspartate receptor ligands including ketamine, amantadine, dextromethorphan (except low dose intermittent use for cough), memantine, methadone, dextropropoxyphene, and/or ketobemidone.
12. Amputations of lower extremities (toe amputation is allowed).
13. Any condition, including serious medical conditions that could interfere with the ability of the subject to participate in the study or could confound study assessments.
14. Subjects who meet the criteria for suicidal intent, plan and/or behavior by scoring 3 or 4 on Questions 2 or 13, or 2 or higher on any Questions 1a (only if 1b is coded YES), 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, or 14 based on the Sheehan - Suicidality Tracking Scale at Visit 1 or Visit 2.

Waivers to the exclusion criteria will NOT be allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Aptinyx Clinical Site, Phoenix, Arizona
  - Aptinyx Clinical Site, Anaheim, California
  - Aptinyx Clinical Site, Fresno, California
  - Aptinyx Clinical Site, Norco, California
  - Aptinyx Clinical Site, Santa Monica, California
  - Aptinyx Clinical Site, Tustin, California
  - Aptinyx Clinical Site, New London, Connecticut
  - Aptinyx Clinical Site, Bradenton, Florida
  - Aptinyx Clinical Site, Brandon, Florida
  - Aptinyx Clinical Site, Fort Myers, Florida
  - Aptinyx Clinical Site, Hallandale, Florida
  - Aptinyx Clinical Site, Jupiter, Florida
  - Aptinyx Clinical Site, Miami, Florida
  - Aptinyx Clinical Site, Ocoee, Florida
  - Aptinyx Clinical Site, Orlando, Florida
  - Aptinyx Clinical Site, Tampa, Florida
  - Aptinyx Clinical Site, West Palm Beach, Florida
  - Aptinyx Clinical Site, Columbus, Georgia
  - Aptinyx Clinical Site, Decatur, Georgia
  - Aptinyx Clinical Site, Meridian, Idaho
  - Aptinyx Clinical Site, Flossmoor, Illinois
  - Aptinyx Clinical Site, Hazelwood, Missouri
  - Aptinyx Clinical Site, Berlin, New Jersey
  - Aptinyx Clinical Site, Rochester, New York
  - Aptinyx Clinical Site, Dayton, Ohio
  - Aptinyx Clinical Site, Knoxville, Tennessee
  - Aptinyx Clinical Site, Memphis, Tennessee
  - Aptinyx Clinical Site, Tullahoma, Tennessee
  - Aptinyx Clinical Site, Austin, Texas
  - Aptinyx Clinical Site, Houston, Texas
  - Aptinyx Clinical Site, Plano, Texas
  - Aptinyx Clinical Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- NYX-2925 200 mg Once Daily (QD): NYX-2925 200 mg PO once daily (QD)
- NYX-2925 50 mg QD: NYX-2925 50 mg PO QD
- NYX-2925 10 mg QD: NYX-2925 10 mg PO QD
- Placebo QD: Placebo PO QD
Period: Overall Study
Arm/Group | NYX-2925 200 mg Once Daily (QD) | NYX-2925 50 mg QD | NYX-2925 10 mg QD | Placebo QD
Started | 75 | 77 | 77 | 72
Completed | 73 | 74 | 72 | 69
Not Completed | 2 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- NYX-2925 200 mg QD: NYX-2925 200 mg PO QD
- NYX-2025 50 mg QD: NYX-2925 50 mg PO QD
- Total: Total of all reporting groups
Arm/Group | NYX-2925 200 mg QD | NYX-2025 50 mg QD | NYX-2925 10 mg QD | Placebo QD | Total
Number analyzed (Participants) | 75 | 77 | 77 | 72 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 57 | 60 | 59 | 233
  >=65 years | 18 | 20 | 17 | 13 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 32 | 37 | 137
  Male | 44 | 40 | 45 | 35 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 27 | 28 | 114
  Not Hispanic or Latino | 45 | 47 | 50 | 44 | 186
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 2 | 2 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 17 | 20 | 18 | 15 | 70
  White | 55 | 53 | 55 | 52 | 215
  More than one race | NA — not collected | NA — not collected | NA — not collected | NA — not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 75 | 77 | 77 | 72 | 301
DPN Disease History (years) [Mean (Standard Deviation); unit: years] — Number of years subject experienced DPN - Lower Extremities
  years | 3.97 (2.723) | 3.46 (2.632) | 3.88 (2.528) | 3.91 (2.373) | 3.8 (2.565)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Average Pain Intensity
Description: Change in the NRS score assessing average pain intensity in the past 24 hours; 0=no pain, 10=worst pain imaginable
Time Frame: From baseline (average of -7 to -1) to Week 4 (average of Days 22 through 28)
Population: All subjects who were included in the safety population, were randomized, and had at least 4 post-baseline daily average pain scores are included in the efficacy population. [mixed effects repeated measures (MMRM)]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NYX-2925 200 mg QD | NYX-2025 50 mg QD | NYX-2925 10 mg QD | Placebo QD
Number analyzed (Participants) | 74 | 77 | 77 | 72
score on a scale | -1.50 (0.19) | -1.61 (0.19) | -1.15 (0.19) | -1.23 (0.19)

2. Secondary Outcome: Numeric Rating Scale (NRS) Average Pain Intensity in Patients Who Did Not Use a Concomitant Medication at Baseline
Description: Change in the NRS score assessing average pain intensity in the past 24 hours for patients who did not use a concomitant medication at baseline; 0=no pain, 10=worst pain imaginable
Time Frame: baseline to week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NYX-2925 200 mg QD | NYX-2025 50 mg QD | NYX-2925 10 mg QD | Placebo QD
Number analyzed (Participants) | 37 | 41 | 35 | 35
score on a scale | -1.55 (0.28) | -1.62 (0.26) | -1.42 (0.29) | -1.03 (0.29)

3. Post Hoc Outcome: Numeric Rating Scale (NRS) Average Pain Intensity in Subjects With DPN >= 4 Years
Description: Change in the NRS score assessing average pain intensity in the past 24 hours in patients with DPN >=4 years; 0=no pain, 10=worst pain imaginable
Time Frame: baseline to week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NYX-2925 200 mg QD | NYX-2025 50 mg QD | NYX-2925 10 mg QD | Placebo QD
Number analyzed (Participants) | 36 | 26 | 32 | 33
score on a scale | -1.19 (0.27) | -1.93 (0.31) | -1.00 (0.29) | -0.72 (0.27)
Statistical Analysis 1: Comparison: NYX-2025 50 mg QD vs Placebo QD; Test type: Other; p = 0.004, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are defined as the start of the event occurring on or after the date of first dispensed study drug (Day 1, Baseline Visit) and before or on the last dose (Week 4). The protocol required adverse events to be followed to resolution of the adverse event.
Arm/Group | NYX-2925 200 mg QD | NYX-2925 50 mg QD | NYX-2925 10 mg QD | Placebo QD
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/77 | 0/77 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/77 | 0/77 | 1/72
Other Adverse Events (participants affected / at risk) | 3/75 | 4/77 | 12/77 | 4/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYX-2925 200 mg QD (N=75) | NYX-2925 50 mg QD (N=77) | NYX-2925 10 mg QD (N=77) | Placebo QD (N=72)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (2) — Cholecystitis, Gallbladder perforation
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NYX-2925 200 mg QD (N=75) | NYX-2925 50 mg QD (N=77) | NYX-2925 10 mg QD (N=77) | Placebo QD (N=72)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03219320/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03219320/SAP_001.pdf